CLINICAL TRIAL: NCT00808184
Title: Pharmacokinetic Study of CPT-11, Raltegravir and Midazolam With Characterisation of UGT1A1 Genotype
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PK01/16/08
Record Dates: First submitted 2008-12-11; First posted 2008-12-15 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2010-04

CONDITIONS: Solid Tumor
Keywords: Histologically or cytologically proven solid tumour for which CPT-11 given by the Folfiri regimen
MeSH Terms: interventions — Irinotecan; Raltegravir Potassium; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPT-11 (Active Comparator)
  Interventions: Drug: CPT-11, Raltegravir (Isentress®), Midazolam

INTERVENTIONS:
Drug: CPT-11, Raltegravir (Isentress®), Midazolam

SUMMARY:
The objectives of this study are:

To correlate pharmacokinetic parameters of raltegravir and midazolam with irinotecan (CPT-11) and its metabolite SN-38.

To correlate the genotype of UGT1A1 of patients receiving CPT-11 chemotherapy with irinotecan and raltegravir pharmacokinetic parameters.

To model pharmacokinetic and pharmacodynamic behaviour of CPT-11 in the study population.

DETAILED DESCRIPTION:
To correlate pharmacokinetic parameters of raltegravir and midazolam with irinotecan (CPT-11) and its metabolite SN-38.

To correlate the genotype of UGT1A1 of patients receiving CPT-11 chemotherapy with irinotecan and raltegravir pharmacokinetic parameters.

To model pharmacokinetic and pharmacodynamic behaviour of CPT-11 in the study population.

VI. Abstract of Research Proposal In no more than 300 words, describe concisely the specific aims, hypotheses, methodology and approach of the application, indicating where appropriate the application's importance to science or medicine. The abstract must be self-contained so that it can serve as a succinct and accurate description of the application when separated from it. Please use lay terms. If this not possible, the technical and medical terms should be explained in simple language. The pharmacokinetic parameters of raltegravir will correlate well with irinotecan (CPT-11) and its metabolite SN-38 and better than midazolam.

Raltegravir pharmacokinetic parameters can be used to predict the genotype of UGT1A1 of patients receiving CPT-11 chemotherapy with irinotecan. Patients who are prescribed the CPT-11 containing regimen FOLFIRI will be selected for the study.

Subjects will then undergo the raltegravir and midazolam test one day before the first dose of their chemotherapy. Pharmacokinetic sampling will occur for these 2 days. The raltegravir and midazolam test will be carried out under fasting conditions (minimum 10 hours). Between 8 to 9 am, one mg of midazolam will be administered intravenously over 30 seconds. At the same time, raltegravir 400 mg will be administered orally with water. Blood samples will be drawn at specified times for pharmacokinetic analysis from a heparinised butterfly needle in the opposite arm.

On the next day, FOLFIRI will be administered as follows:

CPT-11 at 180 mg/m2 in 250 mL Normal Saline over 90 min followed by Leucovorin at 400 mg/m2 in 250 mL Normal Saline over 2 hours followed by 5-Flourouracil 400 mg/m2 IV bolus followed by 5-Flourouracil 2400 mg/m2 over 46 hours. Premedications may be administered as per routine clinical practice. Blood will be taken at specified times for pharmacokinetic analysis. The pharmacokinetic parameters of the raltegravir and midazolam will be compared with the pharmacokinetic parameters of CPT-11 and its metabolite SN-38. Correlation analysis will be performed on the parameters to find the raltegravir or midazolam parameters which correlate best with the CPT-11 and SN-38 parameters. CPT-11 and raltegravir parameters will be correlated with UGT1A1 and other demographic information.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven solid tumour for which CPT-11 given by the Folfiri regimen is indicated and prescribed by the attending physician.
* Age above 21 years.
* Measurable or evaluable disease
* Karnofsky performance status > 70%
* Life expectancy > 3 months
* WBC > 3.0 x 103/?l; ANC > 1500/?l
* Hemoglobin > 9.0 g/dl
* Platelets > 100000/?l
* Creatinine < 1.5 x ULN or calculated creatinine clearance > 40 ml/min
* Total bilirubin < 1.5 x ULN
* SGOT, SGPT < 5 x ULN unless due to disease

Exclusion Criteria:

* Biologic therapy or chemotherapy within 4 weeks. (Six weeks for prior nitrosoureas or mitomycin C).
* Radiation therapy within 4 weeks if > 25% of bone marrow was irradiated.
* Have not received any medications that are known to be metabolised by UGT1A1 within 30 days of the first dose of CPT-11.
* Short gut syndrome or other causes of malabsorption.
* Colony stimulating factors within 2 weeks.
* Women of childbearing potential not practicing birth control. (Note: by means other than oral contraception)
* Pregnant women
* Severe peripheral neuropathy grade 2 or higher.
* Medical or psychiatric conditions which may impair the patient's ability to provide informed consent.
* Hypersensitivity to CPT-11, raltegravir or midazolam/other benzodiazepines.
* Rapidly progressive intracranial or spinal metastatic disease.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Correlate pharmacokinetic parameters of raltegravir and midazolam with irinotecan (CPT-11) and its metabolite SN-38 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Boon Cher Goh, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore

REFERENCES:
- [Background] Atsumi R, Suzuki W, Hakusui H. Identification of the metabolites of irinotecan, a new derivative of camptothecin, in rat bile and its biliary excretion. Xenobiotica. 1991 Sep;21(9):1159-69. doi: 10.3109/00498259109039556. PMID 1788984
- [Background] Gupta E, Mick R, Ramirez J, Wang X, Lestingi TM, Vokes EE, Ratain MJ. Pharmacokinetic and pharmacodynamic evaluation of the topoisomerase inhibitor irinotecan in cancer patients. J Clin Oncol. 1997 Apr;15(4):1502-10. doi: 10.1200/JCO.1997.15.4.1502. PMID 9193346
- [Derived] Lee LS, Seng KY, Wang LZ, Yong WP, Hee KH, Soh TI, Wong A, Cheong PF, Soong R, Sapari NS, Soo R, Fan L, Lee SC, Goh BC. Phenotyping of UGT1A1 Activity Using Raltegravir Predicts Pharmacokinetics and Toxicity of Irinotecan in FOLFIRI. PLoS One. 2016 Jan 25;11(1):e0147681. doi: 10.1371/journal.pone.0147681. eCollection 2016. PMID 26808671